CLINICAL TRIAL: NCT03715569
Title: CNS Infections Effect on the Inner Ear
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Elisa Skovgaard Jensen, Principal Investigator, Nordsjaellands Hospital
Other Study IDs: PM52008
Record Dates: First submitted 2018-06-01; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: CNS Infection; Inner Ear Hearing Loss; Vestibular Abnormality; Inner Ear Inflammation; Hearing Loss, Sensorineural
MeSH Terms: conditions — Central Nervous System Infections; Hearing Loss, Sensorineural; Labyrinth Diseases | interventions — Vestibular Function Tests; Environmental Biomarkers; Audiometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebral fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort with CNS infections: Otoacoustic emissions (OAE), Wide Band Tympanometry (WBT), Vestibular function tests. Audiometry. MOCA, eGOS are cognitive tests.
  Biomarker is a protein found in the inner ear examined in the cerebral fluid.
  Interventions: Diagnostic Test: Vestibular function; Diagnostic Test: OAE/WBT; Diagnostic Test: Biomarker; Diagnostic Test: MOCA, eGOS; Diagnostic Test: Audiometry
- OAE/WBT control: Healthy individuals: Otoacoustic emissions in normal position with head. Otoacoustic emission in different head positions.
  Interventions: Diagnostic Test: OAE/WBT
- OAE/WBT control: Systemic infection: Otoacoustic emission during admission
  Interventions: Diagnostic Test: OAE/WBT
- OAE/WBT control: ICP changes: Otoacoustic emission on patients without an CNS infection before and after elective lumbare puncture with measurement of intracranial pressure (ICP).
  Interventions: Diagnostic Test: OAE/WBT
- Biomarker control: Inner ear biomarkers in patients without CNS infection. Inner ear fluid examination from patients that underwent elective cochlea implantation.
  Interventions: Diagnostic Test: Biomarker

INTERVENTIONS:
Diagnostic Test: Vestibular function — Vhit, Caloric test
  Groups: Cohort with CNS infections
Diagnostic Test: OAE/WBT — Oto acoustic emissions Wide Band Tympanometry
  Groups: Cohort with CNS infections; OAE/WBT control: Healthy individuals; OAE/WBT control: ICP changes; OAE/WBT control: Systemic infection
Diagnostic Test: Biomarker — Biomarker examination
  Groups: Biomarker control; Cohort with CNS infections
Diagnostic Test: MOCA, eGOS — Cognitive tests
  Groups: Cohort with CNS infections
Diagnostic Test: Audiometry — Hearing test
  Groups: Cohort with CNS infections

SUMMARY:
Study on patients with CNS infections.

DETAILED DESCRIPTION:
Aims and objectives:

The present proposal aims to improve the outcome from central nervous system infections (CNS) by improving the understanding of when and why patients develop hearing loss and other neurological sequelae. The investigators will elucidate the temporal development and restitution of a sensorineural hearing loss and will clarify if any therapeutic window exists, where sequelae can be limited.

Also the investigators will investigate if communication between cochlea and cerebrospinal fluid is a window to the intracranial pressure.

Background:

CNS infections remain diseases with high mortality and morbidity. Among survivors from bacterial meningitis, 30 % suffer hearing loss or deafness arising from injury to the inner ear - the cochlea. From previous work it is known that brain inflammation, brain edema and subsequent pressure changes can be transduced to the inner ear due to communication between the cochlea and cerebrospinal fluid (CSF).

The viability of cochlear hair cells can evaluated by non-invasive measurement of otoacoustic (OAE) emissions which are low-intensity sounds from the cochlea (OAE).

Methods and materials:

The investigators will perform repeated measurements of OAE and Wide Band tympanometry (WBT) in all patients admitted with suspicion of a CNS infection. OAE and WBT will be compared to intracranial pressure (ICP) measured during lumbar puncture as well as clinical-, biochemical- and imaging data. An age-matched control group will be included. At discharge and at follow-up patients will receive a neurological, vestibulare examination, cognitive test and a regular hearing test.

Expected outcome and perspectives:

From repeated measures during a course of disease, the investigators will elucidate the development of a hearing loss and clarify if any therapeutic window exists, where sequelae can be limited. This is also an opportunity to assess OAE as a non-invasive measure of intracranial pressure which is believed to be among the clinical complications responsible for a poor outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a CNS infection admitted to the hospital.

Exclusion Criteria:

* Patients with known hearing loss

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with a CNS infection.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Cochlear damage | Day1-90
  Assess the frequency and timely evolution of sensorineural hearing loss by using OAE/WBT and audiometry.

SECONDARY OUTCOMES:
Vestibular function loss | Day 1-90
  Assess the frequency of vestibular function loss by using VHit and Caloic tests.
Identifying biochemical markers in CSF during a CNS infection | Day 1-90
  Identify biomarkers, such as Cochlin, in CSF and assess their ability to predict sequelae.
Cognitive impairment | Day 90
  Assess the frequency and serverity of cognitive impariment by using MOCA scores.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Brandt, MD, Study Director — Department of infectious diseases
Locations (1):
- Hillerød hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No